CLINICAL TRIAL: NCT04281355
Title: Individualized Locoregional Treatment of Initially Biopsy-proven Node-positive Breast Cancer After Primary Systemic Therapy: The EUBREAST-2 INDAX Trial
Brief Title: Individualized Locoregional Treatment of Initially Biopsy-proven Node-positive Breast Cancer After Primary Systemic Therapy
Acronym: INDAX
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jana de Boniface, Sponsor-Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUBREAST-2 INDAX
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomisation A - Intervention (Experimental): In pathologically node-negative patients on axillary staging (TAD, TLNB, SLNB) after primary systemic treatment, no regional radiotherapy is given and no axillary lymph node dissection are performed.
  Interventions: Procedure: Omission of axillary lymph node dissection; Radiation: Omission of regional irradiation
- Randomisation B - Intervention (Experimental): In pathologically node-positive patients on axillary staging (TAD, TLNB, SLNB) after primary systemic treatment, full axillary and regional radiotherapy is given but no axillary lymph node dissection performed.
  Interventions: Procedure: Omission of axillary lymph node dissection

INTERVENTIONS:
Procedure: Omission of axillary lymph node dissection — Axillary lymph node dissection will be replaced by axillary radiotherapy in Randomisation B
Radiation: Omission of regional irradiation — Regional irradiation will be omitted in the interventional arm of Randomisation A.
  Arms: Randomisation A - Intervention

SUMMARY:
In clinically node-positive (cN+) breast cancer, preoperative systemic therapy (PST) is common. With increasing rates of complete tumour eradication, there is a need for de-escalation of locoregional treatment in the interest of decreased morbidity.

In order to individually adapt postoperative therapies, axillary staging is crucial. Axillary lymph node dissection (ALND) comes at a high risk of arm morbidity. There is extreme divergence in the use of less extensive staging methods, i.e. targeted lymph node biopsy (TLNB), sentinel node biopsy (SNB) or both (TAD), and in the use of subsequent locoregional treatment, since prospective data are largely lacking.

The main purpose of the European INDAX trial is to implement de-escalated staging and evaluate which regional treatment, individually adapted to the response after PST, is oncologically safe but least harmful.

Population: cN+ breast cancer patients receiving PST, recruited 2021-2025. Staging by TLNB, TAD or SNB.

Intervention: Negative staging (ypN0, Randomisation A, N=1433): no regional treatment. Positive staging (ypN+, Randomisation B, N=1513): no ALND but regional radiotherapy (rRT).

Control: Randomisation A: rRT only. Randomisation B: ALND plus rRT.

Outcome: Invasive disease-free survival (non-inferiority), arm morbidity and quality of life.

Drug tests in whole-tumour organoid cultures, algorithm-based digital image analysis and gene expression analysis are performed to improve response prediction, facilitate tailoring of PST and increase eradication rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary invasive breast cancer cT1-cT3
* cN1 status prior to PST
* Cytological or histological proof of axillary metastasis before PST
* Full tumour biology available before initiation of PST
* Oral and written consent
* Age ≥ 18 years

Exclusion Criteria:

* Biopsy-confirmed regional nodal metastases outside of the ipsilateral axilla
* Distant metastases at diagnosis
* Inflammatory breast cancer
* Previous axillary surgery
* Previous radiotherapy to ipsilateral breast, chest or axilla
* History of prior invasive breast cancer
* Ongoing pregnancy or breast-feeding
* Bilateral invasive breast cancer
* Medical contraindication for radiotherapy or inability to receive recommended radiotherapy
* Medical contraindication for adjuvant endocrine treatment, if indicated
* Inability to absorb or understand the meaning of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
iDFS | 5 years
  Invasive disease-free survival

IPD SHARING:
Plan to Share IPD: Undecided